CLINICAL TRIAL: NCT01123031
Title: Oral vs Intravenous Proton Pump Inhibitor（PPI） in Patients With Peptic Ulcer Bleeding After Successful Endoscopic Therapy- a Prospective Randomized Comparative Trial
Brief Title: Oral vs Intravenous and Proton Pump Inhibitor (PPI）for Peptic Ulcer Bleeding (PUB)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated and the PI has left the institution.
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCH-100118
Record Dates: First submitted 2010-04-13; First posted 2010-05-14 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Upper Gastrointestinal Bleeding
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Lansoprazole; Esomeprazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- lansoprazole (Active Comparator): lansoprazole 30 mg four times daily for three days followed by 30 mg once daily for two months
  Interventions: Drug: lansoprazole
- esomeprazole (Active Comparator): esomeprazole 160 mg/day continuous infusion for three days followed by 40 mg once daily orally for two months
  Interventions: Drug: esomeprazole

INTERVENTIONS:
Drug: lansoprazole — lansoprazole 30 mg four times daily for three days followed by 30 mg once daily for two months
  Other Names: takeprone
  Arms: lansoprazole
Drug: esomeprazole — esomeprazole 160 mg/day continuous infusion for three days followed by 40 mg once daily orally for two months
  Other Names: nexium
  Arms: esomeprazole

SUMMARY:
A bleeding peptic ulcer remains a serious medical problem with significant morbidity and mortality. Endoscopic therapy significantly reduces further bleeding, surgery, and mortality in patients with bleeding peptic ulcers and is now recommended as the first hemostatic modality for these patients.

In the past few years, adjuvant use of a high-dose proton pump inhibitor (PPI) after endoscopic therapy has been endorsed in some studies. Laine and Javid et al found that oral PPI and IV PPI had a similar intragastric pH response in the past two years. Therefore, whether oral can replace IV in the management of peptic ulcer bleeding is the objective in this study.

The investigators enrolled 130 patients with active bleeding or nonbleeding visible vessels（NBVV） in this study. They are randomly assigned as oral lansoprazole or IV nexium group. All patients receive successful endoscopic therapy with heater probe or hemoclip placement.

In the lansoprazole group (N=65), 30 mg four times daily is given orally for three days. Thereafter, the patients receive 30 mg lansoprazole orally daily for two months. In the nexium group, 160 mg/day continuous infusion is given for three days. Thereafter, the patients receive 40 mg nexium orally daily for two months.

The primary end point is recurrent bleeding before discharge and within 14 days. At day 14, volume of blood transfused, number of surgeries performed, and the mortality rates of the two groups are compared as well.

DETAILED DESCRIPTION:
A bleeding peptic ulcer remains a serious medical problem with significant morbidity and mortality. Endoscopic therapy significantly reduces further bleeding, surgery, and mortality in patients with bleeding peptic ulcers (1) and is now recommended as the first hemostatic modality for these patients (1, 2).

In the past few years, adjuvant use of a high-dose proton pump inhibitor (PPI) after endoscopic therapy has been endorsed in some studies, two consensus statements and two meta-analysis (3-8). To sustain a high intragastric pH, a high dose of omeprazole has been used in previous studies concerning high-risk peptic ulcer bleeding. In our study, the investigators used 40 mg omeprazole intravenous bolus followed by 160 mg/day continuously infusion for three days. The mean intragastric pH rose to 6.0 one hour after the initial bolus of omeprazole in the omeprazole group; it persisted around this value for the rest of the 24 hours.7 The rebleeding rates were much lower in the PPI as compared with H2RA group (Day 3: 0/50 vs 8/50, p<0.01; Day 14: 2/50 vs 12/50, p<0.01) (4).

How about the route of PPI usage? Oral or IV is the preferred route? Laine et al used oral lansoprazole in patients with peptic ulcer bleeding.9 They were randomly assigned to intravenous lansoprazole (90-mg bolus followed by 9-mg/h infusion) or oral lansoprazole (120-mg bolus followed by 30 mg every 3 hours). A pH was recorded for 24 hours. Mean pH rose above 6 after 2-3 hours of intravenous PPI and 3-4 hours of oral PPI. They concluded that frequent oral PPI may be able to replace the currently recommended intravenous bolus plus infusion PPI therapy in patients with bleeding ulcers. In one recent article, Javid et al also proved that there was no significant difference among various PPIs (omeprazole, pantoprazole, and rabeprazole) given through different routes (IV and oral routes) on raising intragastric pH above 6 for 72 h after successful endoscopic hemostasis in bleeding peptic ulcer.10 In our recent study, the investigators have proved that oral rabeprazole and IV omeprazole are equally effective in preventing rebleeding (13/78 in rabeprazole vs 12/78 in omeprazole, p>0.1) in high-risk bleeding peptic ulcers.11 All secondary outcomes between the two groups were similar, including the amount of blood transfusion, hospital stay, need for surgery and mortality.

The objectives of this study are to assess the outcomes of two different regimens of oral lansoprazole vs high dose of intravenous nexium after endoscopic therapy in patients with peptic ulcer bleeding.

ELIGIBILITY:
Inclusion Criteria:

* A peptic ulcer with active bleeding,a non-bleeding visible vessel (NBVV) or an adherent blood clot at the ulcer base is observed within 24 hours of hospital admission

Exclusion Criteria:

* Patients are excluded from the study if they are pregnant,
* Do not obtain initial hemostasis with endoscopic injection of epinephrine
* Do not give written informed consent
* Have bleeding tendency (platelet count <50×109/L,serum prothrombin <30% of normal,or were taking anticoagulants)
* Uremia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2012-03 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Re-bleeding within 14 days in Patients With Peptic Ulcer Bleeding After Successful Endoscopic Therapy | one year
  recurrent bleeding before discharge and within 14 days

SECONDARY OUTCOMES:
hospital stay | one year
  we measure the above item in high risk patients during hospitalization and within one month
volume of blood transfusion | one year
  we measure the above item in high risk patients during hospitalization and within one month
numbers of operation | one year
  we measure the above item in high risk patients during hospitalization and within one month
numbers of death | one year
  we measure the above item in high risk patients during hospitalization and within one month

CONTACTS AND LOCATIONS:
Overall Officials: Hwai J Lin, M.D., Study Chair — Changhua Christian Hospital

REFERENCES:
- [Derived] Yen HH, Yang CW, Su WW, Soon MS, Wu SS, Lin HJ. Oral versus intravenous proton pump inhibitors in preventing re-bleeding for patients with peptic ulcer bleeding after successful endoscopic therapy. BMC Gastroenterol. 2012 Jun 8;12:66. doi: 10.1186/1471-230X-12-66. PMID 22681960